CLINICAL TRIAL: NCT04247191
Title: Examining a Brief Parent Intervention to Reduce College Student Drinking and Consequences
Brief Title: Parent Intervention to Reduce College Student Drinking and Consequences
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Turrisi, Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2R01AA012529-14 (NIH); R01AA012529 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Underage Drinking; Driving Under the Influence; Drinking, Teen; Drinking, College
MeSH Terms: conditions — Underage Drinking; Driving Under the Influence; Alcohol Drinking in College

STUDY DESIGN:
Intervention Model Description: The first group receives the PBI parent intervention; the second group receives the P-Chat intervention; the third group receive the P-Chat+ intervention; and the fourth group is an assessment-only control.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- P-Chat (Experimental): The P-Chat is a brief individually delivered intervention
  Interventions: Behavioral: P-Chat
- PBI (Experimental): The PBI is a handbook developed by the PI to guide parents in discussing underage drinking, behaviors, and consequences with their teens
  Interventions: Behavioral: PBI
- P-Chat+ (Experimental): The P-Chat+ is a combination of the P-Chat and PBI described above.
  Interventions: Behavioral: P-Chat+
- Control (No Intervention): This group will only complete assessments and will not receive any intervention.

INTERVENTIONS:
Behavioral: P-Chat — The P-Chat is a brief individually delivered intervention based on the principles of Motivational Interviewing (MI) and focuses on increasing parents' motivation to reduce permissiveness toward underage alcohol use while reducing defensiveness and barriers to implementing these rules with their teen.
  Arms: P-Chat
Behavioral: PBI — The PBI is currently a model prevention resource at NIAAA's College Alcohol Intervention Matrix and the research was discussed in the most recent Surgeon General's Report as one of the two prevention approaches that met the rigorous criteria to be considered "efficacious". The first section of the PBI provides an introduction to the problem of substance use. The second section focuses on specific skill building strategies that parents can use to improve communication channels with their teen. Third, is a section that addresses peer influence and provides strategies for developing assertiveness. The fourth section is an in-depth discussion of underage drinking, physiological and psychological effects, mixing alcohol with other drugs, motives for why students drink and don't drink, warning signs, risky binge-type drinking, impaired driving, riding with impaired drivers, alcohol and sexual assault, and how to communicate about parents' experiences when they were young.
  Arms: PBI
Behavioral: P-Chat+ — The P-Chat+ is a combination of the P-Chat and PBI described above. Parents in this arm of the study will receive both interventions.
  Arms: P-Chat+

SUMMARY:
College students' alcohol use continues to be a major public health problem. Among the many consequences of this risky behavior are impaired driving and impaired passenger fatalities. Both college health administrators and parents have requested parent-based interventions (PBIs), and parents have demonstrated ample motivation to communicate with their teens. The proposed research will attempt to enhance an existing effective PBI, curb the alarming trends noted in the literature, and move the field forward by conducting a randomized controlled trial testing a modified version of the PBI that includes additional content for parents to establish clear lines of communication around the important topic of permissiveness (referred to as P-Chat).

DETAILED DESCRIPTION:
High-risk drinking and the associated consequences continue to be significant problems among college students. Among the many consequences of this risky behavior are impaired driving and impaired passenger fatalities. These concerns are further magnified by reports showing: 1) younger drivers are overrepresented in fatal crashes involving impaired drivers; 2)~1 in 6 fatalities are passengers (riders with the impaired drivers; RWID); and 3) although over 1.3 million drivers in the U.S. are arrested for impaired driving annually, they only represent 1% of the estimated 121 million self-reported episodes of impaired driving each year. Despite the benefits noted for the PBI, the investigators' recent NIAAA funded research examining parenting throughout college identified associations between specific parenting behaviors and risky drinking and consequences among students that are not adequately addressed. This research revealed several important trends: 1) many parents allow their teens to drink alcohol in an attempt to take the mystery away and provide opportunities to teach them safer drinking practices; 2) this "parental permissiveness" toward underage drinking, even though it was intended to be protective by parents, had the opposite effect and was significantly associated with increased risky drinking and consequences throughout college even when taking into account other critical factors (e.g., peer norms); 3) even small increases in parental permissiveness translated into students experiencing 4-5 more consequences per year; and 4) the effects of this parental permissiveness was not attenuated by other positive parenting behaviors (e.g., communication, monitoring, modeling). In response to these findings and the initial pilot study showing parents were initially reluctant to change their permissiveness when simply provided with the information about how it was associated with risky student drinking, the investigators embarked on a new endeavor in college student parent intervention research. The investigators developed a brief 15-20 minute intervention (P-Chat) that uses principles of Motivational Interviewing (MI) to reduce defensiveness and modify parents' motives (and behaviors) to change parental permissiveness, and in turn, reduce students' risky drinking and consequences. The investigators have also conducted a pilot randomized controlled trial (RCT) study to demonstrate ability to implement the P-Chat with fidelity; modify parents' willingness to change; and change parents' permissive behaviors. The pilot data provides evidence that the P-Chat intervention has the potential to substantially improve the public health impact of PBIs. The proposed research will examine the P-Chat as a stand-alone intervention and also as an add-on in combination with the original PBI to evaluate the best practice for implementation in a RCT using a rigorous study design.

The primary design is a four-arm randomized control trial with 4 waves of data collection (P-Chat, P-Chat+, PBI Only, and assessment only control). The study will enroll an ethnically diverse sample of 900 parent-student dyads. Students will complete assessments of all the primary, secondary, and tertiary outcomes at four times: pre-intervention baseline and 3-month, 6-month, and 9-month follow-ups. To maximize the diversity of the sample, the investigators are oversampling for 30% racial/ethnic minorities, free of sample bias.

The continuation of the study is to assess the long-term effects of the parent interventions in the 4th (senior) year of college and one year later. Student participants will complete assessments twice: once during their senior year of college and once one year later after transitioning from college. Assessments will include online survey and the Alcohol Use Disorder (AUD) module of the Structured Clinical Interview for DSM-5 (SCID-5) interview at both time points.

ELIGIBILITY:
Inclusion Criteria:

* Parent and teen both consent and complete baseline (forming a dyad testing unit);

Exclusion Criteria:

* Outside of the teen age range; both parent and teen do not consent and complete baseline

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2061 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Examine Changes in Alcohol Use | Baseline, 3 month, 6 month, 9 month, senior year college, 1-year post-college
  A standard drink definition will be provided, indicating that a standard drink consists of 12 oz. of beer or wine cooler, 8.5 oz. of malt liquor, 4 oz. of wine, or 1.5 oz. of hard liquor. Using the Timeline Followback (TLFB; Sobell & Sobell, 1996) participants will indicate how many drinks they consumed on each day of the past three months. For days alcohol was consumed, participants will also note the number of hours spent drinking.
Examine Changes in Consequences of Alcohol Use | Senior year college, 1-year post-college
  Alcohol-related consequences (e.g., said or done embarrassing things, blackout) from the past three months will be measured using the established Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ; Read, Kahler, Strong, & Colder, 2006). Response options will be measured on a 7-point scale ranging from (0) no, not in the past year to (6) 11 or more times in the past year.
Past year Alcohol Use Disorder (AUD) | Senior year college, 1-year post-college
  Past year alcohol use disorder (AUD) will be assessed using the AUD module of the Structured Clinical Interview for DSM-5.

SECONDARY OUTCOMES:
Examine Changes in Impaired Driving (IMPD) Behaviors | Baseline, 3 month, 6 month, 9 month
  Using the TLFB calendar, participants will indicate whether they drove a vehicle after using alcohol(Yes/No).
Examine Changes in Riding with Impaired Driver (RWID) Behaviors | Baseline, 3 month, 6 month, 9 month
  Using the TLFB calendar, participants will indicate whether they rode in a vehicle with a driver that had been drinking (Yes/No).
Examine Changes in Consequences of Alcohol Use | Baseline, 3 month, 6 month, 9 month
  Alcohol-related consequences (e.g., said or done embarrassing things, blackout) from the past three months will be measured using the established Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ; Read, Kahler, Strong, & Colder, 2006). Response options will be measured on a 7-point scale ranging from (0) no, not in the past year to (6) 11 or more times in the past year.

OTHER OUTCOMES:
Examine Changes in Parental Rules about Underage Drinking (Permissiveness) | Baseline, 3 month, 6 month, 9 month
  Adapted from measures by Van Der Vorst et al. (2006), parental permissiveness of underage drinking will be assessed using six items (e.g., I am allowed to drink alcohol on special occasions), based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Parental Communication | Baseline, 3 month, 6 month, 9 month
  Parental communication about alcohol use, IMPD, and RWID will be assessed separately for mothers and fathers. Participants will be asked whether their parent discussed these topics (yes/no) with them within the past three months. Items include topics such as "the importance of not being pressured to drink to fit it" and "the health reasons why you should not be allowed to get drunk once in a while".
Examine Changes in Parental Communications | Baseline, 3 month, 6 month, 9 month
  General Communication (e.g., my mother/father is there for me when I want to talk) will be assessed separately for mothers and fathers based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Alcohol Use Motives | Baseline, 3 month, 6 month, 9 month
  Motives will be assessed for using alcohol (e.g., to be sociable; Cooper, 1994). Responses will be recorded using 5-point scale ranging from (1) almost never/never to (5) almost always/always.
Examine Changes in Alcohol Use Expectancies | Baseline, 3 month, 6 month, 9 month, 12 month
  Expectancies for using alcohol (e.g., I will feel badly about myself because of my drinking) will be measured. Responses will be recorded using 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Willingness to Drink Alcohol | Baseline, 3 month, 6 month, 9 month
  Response options for willingness items will be on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree. Willingness to drink will be measured with three items assessing participants' willingness to 1) drink 1-2 drinks in 2 hours; 2) drink 3-4 drinks in 2 hours; 3) drink 5+ drinks in 2 hours.
Examine Changes in Peer Descriptive Norms | Baseline, 3 month, 6 month, 9 month
  Perceived peer descriptive norms of drinking will be measured using the Daily Drinking Questionnaire (DDQ; Collins, Parks, & Marlatt, 1985) by assessing how much alcohol, on average, participants' closest friends drink each day of the week.
Examine Changes in General Parental Practices | Baseline, 3 month, 6 month, 9 month
  General Parenting Practices (e.g., if I had a personal problem I could ask my mother/father for help) will be assessed separately for mothers and fathers based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Peer Injunctive Norms | Baseline, 3 month, 6 month, 9 month
  Perceived peer injunctive norms will be measured by indicating the level of approval participants' closest friends would have from a list of items (e.g., drinking alcohol every weekend) on a 7-point scale ranging from (1) strongly disapprove to (7) strongly approve.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Turrisi, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No